CLINICAL TRIAL: NCT00544063
Title: Phase I Study Evaluating the Feasibility of Chemotherapy With Capecitabine, Irinotecan, and Oxaliplatin in Patients With Metastatic Carcinoma
Brief Title: Capecitabine, Irinotecan, and Oxaliplatin in Treating Patients With Metastatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000564073; CLCC-XEL-IRIN-OX; INCA-RECF0416; VA-XIOX; EudraCT-2005-004567-38
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan; Oxaliplatin

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, irinotecan, and oxaliplatin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of capecitabine when given together with irinotecan and oxaliplatin in treating patients with metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicities of capecitabine.

Secondary

* Determine the recommended phase II dose of capecitabine.
* Define the toxicity profile.
* Evaluate potential antitumor activity in terms of objective response, duration of response, and time to disease progression.
* Evaluate the pharmacokinetic profile of capecitabine and irinotecan hydrochloride.

OUTLINE: This is a dose-escalation study of capecitabine conducted in two parts.

* Part I: Patients receive irinotecan hydrochloride IV over 90 minutes on day 1 and oral capecitabine twice daily on days 1-7. Treatment repeats every 2 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity.

Cohorts of up to 6 patients receive escalating doses (up to 5 dosages) of capecitabine. The maximum tolerated dose (MTD) is defined as the dose at which 50% of patients experience toxicity during the first 2 courses of therapy.

* Part II: Patients receive oxaliplatin IV over 2 hours and irinotecan hydrochloride IV over 90 minutes on day 1 and oral capecitabine on days 1-7. Treatment repeats every 2 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity.

Cohorts of up to 6 patients receive escalating doses (up to 7 dosages) of capecitabine. The MTD is defined as in part I.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed metastatic carcinoma

  * Primary tumor may be present
  * No curative therapy available or the patient achieved no response to prior standard therapy
  * Nonresectable metastatic disease
* Measurable, evaluable, or nonevaluable disease

Exclusion criteria:

* Symptomatic brain metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin < 1.25 times upper limit of normal (ULN) (1.5 times ULN if due to liver metastases)
* Transaminases < 3 times ULN (5 times ULN if due to liver metastases)
* Alkaline phosphatase ≤ 3 times ULN
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance > 30 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception

Exclusion criteria:

* Severe concurrent infection or major organ failure, including any of the following:

  * Cardiac disease
  * Diabetic decompensation
  * Clinically active infection
* Prior severe toxicity from fluorouracil
* Intestinal obstruction or subobstruction
* Malabsorption syndrome
* Peripheral neuropathy
* Uncontrolled epilepsy

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* At least 4-6 weeks since prior anticancer chemotherapy

Exclusions criteria:

* Prior chemotherapy with any of the study drugs
* Prior major intestinal resection
* Concurrent participation in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of capecitabine
Dose-limiting toxicities

SECONDARY OUTCOMES:
Recommended phase II dose of capecitabine
Toxicity profile
Objective response
Duration of response
Time to disease progression
Pharmacokinetic profile of capecitabine and irinotecan hydrochloride

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ychou, MD, PhD — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France